CLINICAL TRIAL: NCT04303234
Title: Intraoperative Pain During Restorative Treatment Of Maxillary First Permanent Molars Using Artinibsa Versus Artpharma In Children After Infiltration Technique: A Randomized Clinical Trial
Brief Title: Assess Intraoperative Pain for Restorative Treatment of Maxillary 1st Permanent Molars Using Artinibsa Versus Artpharma in Children During Infiltration Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amani Hamed Hashem AL-Aidaros, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2020-03-08
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Pain
Keywords: Articaine; Infiltration technique; Restoration primary teeth; Intraoperative pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: single ( participant ) because the two interventions used in this trial are easily recognized by the investigator but the participant and the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artinibsa (Active Comparator): Powerful local anesthetic with short time for patients who can not tolerate normal doses of vasoconstrictor latency.
  High lipid solubility gives a better diffusion through the soft tissue and bone being very effective in infiltrative techniques.
  Duration:
  Latency time: 2 minutes
  Each mL contains:
  4%Articaine 1:100000. Hydrochloride 40.00 mg, Epinephrine (D.C.I) 0.005 mg tartrate
  Interventions: Other: Artinibsa
- Artpharma (Experimental): Its a special amide local anesthetic contain 4% articaine with epinephrine 1/200000 as a vasoconstrictor ,Contains only sulfite as a stabilizer (max 0.31 mg)
  Interventions: Other: Artpharma

INTERVENTIONS:
Other: Artinibsa — local anaesthetic solution with a short latency time. Its high lipid solubility gives it better diffusion through soft tissues and bone and makes it highly effective for infiltrative techniques.Each ml contains 4%Articaine 1:100000.
  Arms: Artinibsa
Other: Artpharma — Its a special amide local anesthetic contain 4% articaine with epinephrine 1/200000 as a vasoconstrictor ,Contains only sulfite as a stabilizer (max 0.31 mg)
  Arms: Artpharma

SUMMARY:
The aim of this study is to assess Intraoperative pain for restorative treatment of Maxillary First Permanent Molars using Artinibsa Versus Artpharma in children during infiltration technique.

DETAILED DESCRIPTION:
Local anesthesia is very important during dental procedure because it's a temporary loss of sensation which will lead to decrease the pain. Local anesthesia started with discovery of Cocaine in 1860. Followed by developments of Novocaine 1904 and lignocaine in 1942 by Lofgren. It became the gold standard drug compared to other local anesthetic. Later, several new drugs were discovered such as:Bupivacaine, Articaine, Mepivicaine etc. Articaine Hydrochloride (HCL) was available in Germany since 1976. It's the only amide local anesthesia containing ester group in its molecular structure leading to metabolizing of the drug by both plasma esterases and liver microsomal enzymes, the clinical efficacy and advantages of articaine is the duration of its anesthetic effect and its superior diffusion through the bony tissue.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-10 years old
* Mentally capable of communication
* Cooperative children need restorative treatment

Exclusion Criteria:

* Medically compromised patient
* Primary teeth requiring pulpotomy or pulpectomy
* Parent or guardians who refuse participating in the study

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — 8-10 years old
Enrollment: 46 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Pain: Wong Baker rating scale | During the procedure.
  Measuring by using Wong Baker rating scale the measuring unite is :Scale (0-10) including six faces.

SECONDARY OUTCOMES:
Onset of anesthesia | Immediately after the injection.
  is measuring by using stop watch and the unite is minutes. the unit is : minutes
The sensation after injection | Immediately after the injection.
  Evaluating the effect of the anesthesia by checking mucosa using the probe and measuring unite is binary (Yes or No)
Time of numbness disappear | 2 hours postoperatively after the procedure.
  Time of disappearance of numbness sensation by asking the parent/child and measuring is binary (Yes or No).

IPD SHARING:
Plan to Share IPD: No